CLINICAL TRIAL: NCT00005290
Title: Epidemiology of Interstitial Lung Disease
Status: Terminated | Type: Observational
Why Stopped: Not a clinical trial & was inadvertently entered into the system.
Sponsor: University of New Mexico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2012; R01HL040587 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lung Diseases; Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Interstitial

SUMMARY:
To establish a population-based registry of interstitial lung disease in Bernalillo County, New Mexico.

DETAILED DESCRIPTION:
BACKGROUND:

Although many investigations have been conducted to characterize the pathogenesis of interstitial lung diseases, few examined the epidemiology of these disorders in a general population. The establishment of the registry represented the first step in a sequence of investigations designed to characterize the epidemiology of the interstitial lung diseases. The registry initially served a descriptive purpose; the incidence of the interstitial lung diseases was measured in a defined population. Subsequently the registry served as a mechanism for ascertaining cases for a case-control study. Finally, the registry provided population-based data for clinical purposes on presentation, physiology, and natural history of the interstitial lung diseases.

DESIGN NARRATIVE:

The resources of the New Mexico Tumor Registry were adapted to identify new cases of interstitial lung disease in Bernalillo County. Other sources of information for identifying new cases included pulmonary physicians, primary care physicians, death certificates, and autopsies. After a case of interstitial lung disease had been identified from the various sources of information, data collection included an interviewer-administered symptoms questionnaire, abstracted medical record data, phlebotomy for measurement of serum precipitins, and evaluation of available chest x-rays and biopsy materials. Follow-up was used to determine the natural history of the disease.

The study was renewed in 1993 to complete the work conducted from 1988 through 1992. Case-ascertainment, data collection, and follow-up of incident cases of ILD identified during the period 10/1/88-9/30/92 were completed. The incidence of ILDs was described. The clinical characteristics of patients with ILDs were described. The prognosis of the most common ILDs were described.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-04; Study Completion 1997-06

REFERENCES:
- [Background] Mapel DW, Samet JM, Coultas DB. Corticosteroids and the treatment of idiopathic pulmonary fibrosis. Past, present, and future. Chest. 1996 Oct;110(4):1058-67. doi: 10.1378/chest.110.4.1058. No abstract available. PMID 8874268
- [Background] Coultas DB, Hughes MP. Accuracy of mortality data for interstitial lung diseases in New Mexico, USA. Thorax. 1996 Jul;51(7):717-20. doi: 10.1136/thx.51.7.717. PMID 8882079
- [Background] Coultas DB, Zumwalt RE, Black WC, Sobonya RE. The epidemiology of interstitial lung diseases. Am J Respir Crit Care Med. 1994 Oct;150(4):967-72. doi: 10.1164/ajrccm.150.4.7921471.
- [Background] Mulloy KB, Coultas DB, Samet JM. Use of chest radiographs in epidemiological investigations of pneumoconioses. Br J Ind Med. 1993 Mar;50(3):273-5. doi: 10.1136/oem.50.3.273. PMID 8457495
- [Background] Mapel DW, Hunt WC, Utton R, Baumgartner KB, Samet JM, Coultas DB. Idiopathic pulmonary fibrosis: survival in population based and hospital based cohorts. Thorax. 1998 Jun;53(6):469-76. doi: 10.1136/thx.53.6.469. PMID 9713446